CLINICAL TRIAL: NCT00708422
Title: Examination of Ocular Surface Effects With Administration of TRAVATAN Z® and Xalatan®
Brief Title: Effects of Travatan Z and Xalatan on Ocular Surface Health
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMA-08-07
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Ocular surface health; OSDI; TFBUT; Glaucoma; Ocular hypertension; Corneal staining
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost (Experimental): One drop self-administered in the study eye(s) once daily at night for 12 weeks
  Interventions: Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®)
- Latanoprost (Active Comparator): One drop self-administered in the study eye(s) once daily at night for 12 weeks
  Interventions: Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®)

INTERVENTIONS:
Drug: Travoprost ophthalmic solution 0.004% with SofZia® preservative system (TRAVATAN Z®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 12 weeks (84 days). Referred to as travoprost.
  Other Names: TRAVATAN Z®; travoprost
  Arms: Travoprost
Drug: Latanoprost ophthalmic solution 0.005% (XALATAN®) — Ophthalmic solution for the treatment of open-angle glaucoma or ocular hypertension, one drop a day, dosed topically for 12 weeks (84 days). Referred to as latanoprost.
  Other Names: XALATAN®; latanoprost
  Arms: Latanoprost

SUMMARY:
The purpose of this randomized, double-masked, parallel-group, multicenter study is to evaluate ocular surface effects after the administration of travoprost with SofZia® preservative system or Xalatan once daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of primary open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion) or ocular hypertension in at least one eye (study eye).
* Use of BAK (benzalkonium chloride) containing intraocular pressure (IOP) lowering medication for a minimum of one year, including latanoprost (Xalatan®) monotherapy for at least 6 months prior to Visit 1.
* IOP controllable and stable on the study medication alone (both eyes).
* Believed to have ocular surface disease (OSD).
* Tear Break-up Time (TBUT) of ≤ 6 seconds in the study eye.
* Willing and able to discontinue the use of any topical ocular medication other than the study medication or BAK free artificial tears for the duration of the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Current use or use within the last 3 months of cyclosporine ophthalmic emulsion 0.05% (Restasis®), topical ocular steroids, or topical ocular non-steroidal anti-inflammatory drugs.
* Current use of punctual plugs.
* Women of childbearing potential not using reliable means of birth control.
* Women who are pregnant or lactating.
* Suspected or diagnosed with Sjogrens's syndrome.
* Current use of any brand of artificial tears containing BAK.
* Use of any systemic medications on a chronic basis not on a stable dosing regimen for at least 30 days prior to Visit 1, or an anticipated change in dosing regimen of medications during the course of the study.
* Intraocular conventional surgery or laser surgery in study eyes less than six months prior to Visit 1.
* Current use of contact lenses within 30 days of Visit 1.
* Participation in any other investigational study within 30 days prior to Visit 1.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Vittitoe, RN, MPH, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 21 US study centers. Eligible patients having a diagnosis of open-angle glaucoma or ocular hypertension and abnormal TBUT were enrolled.
Pre-assignment Details: 231 patients were enrolled in the study and evaluated for safety. Baseline characteristics are presented for all patients who received the test article and completed the study (intent-to-treat): 226.
Groups:
- Travoprost: One drop self administered in the study eye(s) once daily at night for 12 weeks
Period: Overall Study
Arm/Group | Travoprost | Latanoprost
Started | 116 | 115
Completed | 112 | 114
Not Completed | 4 | 1
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost | Latanoprost | Total
Number analyzed (Participants) | 112 | 114 | 226
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 44 | 78
  >=65 years | 78 | 70 | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 66 | 140
  Male | 38 | 48 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Change at 12 Weeks (Day 84) From Baseline (Day 0) in Tear Film Break Up Time (TBUT)
Description: Tear film break-up time was assessed by the same examiner both visits using the same slitlamp/settings. Examiner instilled fluorescein onto the patient's eye, after which the patient blinked several times, then kept the eye open. Immediately thereafter, the examiner used a stopwatch to time the occurrence of the first break in the fluorescein film. Three consecutive measurements were taken and averaged for actual TBUT. TBUT at Baseline (Day 0) was subtracted from TBUT at 12 weeks (Day 84) and reported as change. A higher number represents a lengthening in the tear film break up time.
Time Frame: 12 weeks (Day 84)
Population: Intent-to-treat: All patients who received test article and completed the trial.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 112 | 113
seconds | 0.8 (1.5) | 1.1 (2.7)

2. Secondary Outcome: Mean Change at 12 Weeks (Day 84) From Baseline (Day 0) in Ocular Surface Disease Index (OSDI) Score
Description: The OSDI is a 12-question validated questionnaire (resultant overall 0-100 score) used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision, where 0 = normal and 100 = severe. The OSDI questionnaire was administered at both visits and completed by the patient with no assistance from the office staff, physician, or anyone else. The baseline OSDI score was subtracted from the 12-week OSDI score and reported as change. A negative number represents a perceived improvement in ocular health.
Time Frame: 12 weeks (Day 84)
Population: Intent-to-treat: All patients who received test article and completed the trial.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Travoprost | Latanoprost
Number analyzed (Participants) | 112 | 112
Units on a scale | -0.0 (11.4) | -1.3 (16.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 11 July 2008 through 03 August 2009.
Description: Patients were queried about any symptoms they may have experienced that would suggest an AE by asking, "Since your last visit, have you had any health problems?" This reporting group includes all patients who received test article.
Arm/Group | Travoprost | Latanoprost
Serious Adverse Events (participants affected / at risk) | 1/116 | 1/115
Other Adverse Events (participants affected / at risk) | 0/116 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Travoprost (N=116) | Latanoprost (N=115)
Cellulitis (Infections and infestations) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The subjective nature of the OSDI may not be sensitive enough to detect the effects of preservatives on the corneal surface. The measurement and quantification of OSD remains a considerable clinical challenge (Pflugfelder and Baudoin, 2011).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.